CLINICAL TRIAL: NCT05120908
Title: Social Isolation and Discrimination as Stressors Influencing BGM Alterations
Brief Title: Discrimination and the Brain-Gut-Microbiome (BGM) Axis
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Arpana Church, Associate Professor, University of California, Los Angeles
Other Study IDs: IRB # 20-002326
Record Dates: First submitted 2021-10-21; First posted 2021-11-16 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Discrimination, Racial; Social Isolation; Stress
Keywords: Obese; Mexican Women; Filipina Women; Overweight; Brain-Gut Microbiome; MRI; Metabolome
MeSH Terms: conditions — Racism; Social Isolation; Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool and plasma are collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mexican Women: Mexican, premenopausal women ages 18-50.
- Filipina Women: Filipina, premenopausal women ages 18-50.

SUMMARY:
Obesity is a major public health problem related to a variety of illnesses such as heart disease and diabetes. Prior research indicates that social stressors contribute to risk for obesity, possibly through alterations in diet and physical activity. However, it is not fully clear how these alterations contribute to obesity. The purpose of this study is to examine how the stressors of social isolation and discrimination relate to eating behaviors and dietary patterns, and further, how these behaviors affect the brain-gut-microbiome (BGM) connections. This study will focus on Mexican and Filipina women because research shows that they encounter a high burden of obesity and exposure to social stressors. Approximately 300 Mexican and Filipina women will be screened and enrolled. They will then provide information about social stressors via food diaries, physical body measures (e.g. waist circumference), questionnaire data regarding diet and eating behaviors, and measures of physical activity. Stool and serum will be collected to analyze microbes and metabolomics, and MRI to assess brain changes in the reward network. Analytic techniques will be used to integrate data from these multiple data sources. This analysis will determine the unique differences associated with ethnicity and social stressors in moderating eating behaviors and dietary patterns. The results of this study will provide new information about a possible pathway whereby social stressors affect behavioral, neurological and microbiome mechanisms related to obesity risk and provide new information in BGM patterns in two understudied ethnic groups. In the long term, this research may suggest possible approaches for intervention that may help reduce inequalities in obesity and related health problems.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal females
* Ages 18-50
* Mexican or Filipino ancestry
* BMI 19-40
* Fluent in English
* Right-handed

Exclusion Criteria:

Co-Morbidities including but not limited to:

* Type I diabetes (insulin dependent)
* Vascular disease
* Drastic weight loss (more than 10lbs over the preceding 2months)
* Frequent Strenuous exercise (i.e. marathon runners/heavy weight lifting)
* Abdominal surgeries including weight loss surgery, or partial/complete resection of the stomach or bowel
* Untreated thyroid disease
* Neurological disease
* Major medical condition that may put the subject at risk or interfere with data collection as determined by the PI/MD
* Chronic pain
* Diagnosed DSM IV active psychiatric illness including eating disorders. Must not be active or present for at least 2 years.
* Use of medications known to affect hunger, satiety, and/or appetite.
* Unable to safely participate in the MRI (claustrophobia, presence of devices affected by MRI such as pacemakers, neurostimulators, or any metallic foreign body, etc.)
* Pregnant, lactating, postpartum less than 6mo
* Women of childbearing age who are not practicing birth control or are planning to get pregnant during the study.
* Body weight at enrollment greater than 400lbs due to weight restrictions on the MRI table
* Use of oral/IV antibiotics within the last 3 months
* Use of probiotics in the last month
* Heavy use of tobacco, alcohol, and/or drug use/abuse
* Significant change in usual diet and/or weight loss of more than 10lbs in the last 2months
* Refugees or recent immigration of less than 2 years in the USA.
* Temporary workers/visitors/students
* Recent international travel if more than 3 weeks within the last 3 months.

Use of the following medications is exclusionary:

* Opiates/narcotics
* Chronic daily use of high dose OTC analgesics
* Anti-seizure medications
* Medications for appetite suppression
* Chronic use of laxatives/antidiarrheals, medications affecting GI motility
* Insulin
* Bile Acid Sequestrants
* Centrally acting medications that will interfere with the neuroimaging testing
* Thyroid replacement medications (OK if stable for at least 3mo)
* Heavy use of tobacco/cannabis
* Heavy use of alcohol ( >7/week for women)
* Antidepressants (5HT3's/Tricyclics) (OK if stable for at least 3mo)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants recruited from the greater Los Angeles Mexican & Filipina female population.
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Multimodal Brain Signatures | Measured once at Visit 2. Scan lasts about 1.5 hour.
  Neuroimaging of participants brain via MRI procedure.
Microbiome - Stool | Collected twice by the participant at home between Visit 1 and Visit 2, lasting no more than 2 weeks after the first appointment.
  Measurement of 16S RNA, shotgun metagenomics, and metabolomics via stool specimen.
Microbiome - Blood | Collected once at Day1.
  Measurement of 16S RNA, shotgun metagenomics, and metabolomics via blood specimen.

SECONDARY OUTCOMES:
Systolic and Diastolic Blood Pressure | Measured once at Day 1.
  Measurement of the pressure of circulating blood at rest.
Questionnaire Data - Diet | Self-reported by the participant at home between Visit 1 and Visit 2, lasting no more than 2 weeks after the first appointment.
  Use of validated surveys including the Food Frequency questionnaire, Food choice questionnaire.
Questionnaire Data - Stressors | Self-reported by the participant at home between Visit 1 and Visit 2, lasting no more than 2 weeks after the first appointment.
  Use of validated surveys including, Social isolation scale, Social network engagement, Family cohesion, Acculturative stress, Perceived stress scale, Everyday Discrimination, and major discrimination.
Anthropometrics - waist & hip circumference | Measured once at Day 1.
  Measurement of waist and hip circumference(cm).
Anthropometrics - BMI | Measured once at Day 1.
  Measurement of height(in) and weight(lbs), used to calculate BMI.
Questionnaire Data - Physical Activity | Self-reported by the participant at home between Visit 1 and Visit 2, lasting no more than 2 weeks after the first appointment.
  Use of validated surveys including the international physical activity questionnaire.
Questionnaire Data - Health | Self-reported by the participant at home between Visit 1 and Visit 2, lasting no more than 2 weeks after the first appointment.
  Use of validated surveys including the health eating index.
Questionnaire Data - Ingestive Behaviors | Self-reported by the participant at home between Visit 1 and Visit 2, lasting no more than 2 weeks after the first appointment.
  Use of validated surveys including the Yale food addiction scale, Three-Factor Eating questionnaire, Reward-based eating drive, General food craving questionnaire - trait-reduced, Cravings and Want to eat Assessments to food cues.

OTHER OUTCOMES:
Differences in Multimodal Brain Signatures | Measured at optional follow up visit at 3 and/or 6 month mark. Scan lasts about 1.5 hour.
  Neuroimaging of participants brain via MRI procedure.
Differences in Microbiome - Stool | Collected twice by the participant at home before the 3 and/or 6 month follow up appointment, occurring approximately 3 and 6 months after the second (MRI) appointment.
  Measurement of 16S RNA, shotgun metagenomics, and metabolomics via stool specimen.
Differences in Microbiome - Blood | Collected once at the 3 and/or 6month follow up appointment, occurring approximately 3 and 6months after the second (MRI) appointment.
  Measurement of 16S RNA, shotgun metagenomics, and metabolomics via blood specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Arpana Gupta, PhD, Principal Investigator — The Regents of the University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
At this time there is no plan to make the de-identified data available for sharing with other researchers.